CLINICAL TRIAL: NCT01045317
Title: An Exploratory, Open Label, Randomized, Parallel Group Study To Investigate The Pharmacokinetics Of Single Intravenous And Oral Micro Doses Of [14-C]-PF-04776548 In Healthy Male Subjects
Brief Title: A Study To Investigate The Clearance Of PF-04776548 From The Body Following A Very Low (Micro) Dose Of The Compound Using A Low Level Of Radiotracer To Help Quantify Expected Low Concentrations Of PF-04776548 In The Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: B1711001
Record Dates: First submitted 2010-01-08; First posted 2010-01-11 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2010-04

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: micro-dose; pharmacokinetics; open label; PF-04776548
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intravenous or oral administration (Experimental)
  Interventions: Drug: PF-04776548

INTERVENTIONS:
Drug: PF-04776548 — single intravenous or oral administration of 0.1mg PF-04776548.

SUMMARY:
To investigate the pharmacokinetics of PF-04776548 following administration of a micro-dose of PF-04776548 via both intravenous and oral routes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 65 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests).
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 21 drinks/week (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) within 6 months of screening.
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: For IV dosing: Cmax, Tmax, AUClast, AUCinf, t½, CL, Vss. For oral dosing: Cmax, Tmax, Tlag, AUClast, AUCinf, t½, CL/F, Vz/F, F. | 14 days

SECONDARY OUTCOMES:
Safety and toleration: adverse events will also be reported. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Ruddington Fields, Nottingham, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1711001&StudyName=A%20Study%20To%20Investigate%20The%20Clearance%20Of%20PF-04776548%20From%20The%20Body%20Following%20A%20Very%20Low%20%28Micro%29%20Dose%20Of%20The%20Compound%20Using%20A%20Lo